CLINICAL TRIAL: NCT03190369
Title: A 26-week, Multicenter, Double-blind, Randomized, Placebo-controlled Parallel Group Study to Evaluate the Efficacy and Safety of a Single Dose of 6 mL of Hylan G-F 20 (Synvisc-One®) in Chinese Patients With Symptomatic Osteoarthritis of the Knee
Brief Title: Randomized Study of the Efficacy and Safety of a Single Dose of Synvisc-One® in Chinese Patients With Symptomatic Osteoarthritis of the Knee
Acronym: C-SOUND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC12723; U1111-1131-0507 (Other: UTN)
Record Dates: First submitted 2017-06-14; First posted 2017-06-16 (Actual); Results first posted 2020-02-05 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants received a single IA injection of phosphate buffered saline on Day 1 and were observed for 26 weeks.
  Interventions: Drug: Placebo
- Hylan G-F 20 (Experimental): Participants received a single IA injection of 6 mL Hylan G-F 20 (Synvisc-One) on Day 1 and were observed for 26 weeks.
  Interventions: Device: Hylan G-F 20 (GZ402662/SAR402662)

INTERVENTIONS:
Device: Hylan G-F 20 (GZ402662/SAR402662) — Pharmaceutical form: Solution for injection
  Route of administration: Intra articular
  Other Names: Synvisc-One
  Arms: Hylan G-F 20
Drug: Placebo — Pharmaceutical form: Solution for injection
  Route of administration: Intra articular
  Arms: Placebo

SUMMARY:
Primary Objective:

-To evaluate the efficacy of a single 6-milliliter (mL) intra-articular (IA) injection of Hylan G-F 20 measured by Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Numerical Rating Scale (NRS) 3.1 A1 score, in comparison to an IA placebo injection over 26 weeks, in Chinese participants with symptomatic Osteoarthritis (OA) of the knee.

Secondary Objectives:

* To evaluate the efficacy of a single 6-mL IA injection of Hylan G-F 20 measured by 7-day average score of WOMAC A1 pain sub-score in comparison to an IA placebo injection over 26 weeks.
* To evaluate the efficacy of a single 6-mL IA injection of Hylan G-F 20 measured by WOMAC A, patient global assessment (PTGA) and clinical observer global assessment (COGA) in comparison to an IA placebo injection over 26 weeks.
* To evaluate the response rate of a single 6-mL IA injection of Hylan G-F 20 in comparison to an IA placebo injection over 26 weeks. Response was defined as WOMAC A1 greater than or equal to (>=) 2-point improvement from baseline on NRS.
* To evaluate the safety of a single 6-mL IA injection of Hylan G-F 20, in comparison to an IA placebo injection over 26 weeks.

DETAILED DESCRIPTION:
The duration of the study was 29 weeks at maximum. The screening and wash-out period lasted for up to 14 days, depending on the half-life of the medications followed by an 8-day baseline period including the treatment day. Overall, there were up to 21 days between signing informed consent (at screening visit) and the randomization (Day 1). Treatment was administered on Day 1, and follow-up period was 26 weeks.

ELIGIBILITY:
Inclusion criteria :

* Symptomatic OA of the target knee joint with WOMAC A1 NRS score of >=4.0 and less than or equal to (<=) 8.0 as recorded in the baseline period.
* Confirmed by standard X-rays performed within 3 months prior to screening visit: modified Kellgren-Lawrence Numerical Grading System of Grade I-III in the target knee joint.
* According to the American College of Rheumatology (ACR) Criteria.
* With failure to respond adequately to conservative non-pharmacologic therapy and/or simple analgesics, such as acetaminophen.
* Participant was willing and was able to provide signed informed consent prior to any study related procedures being performed.

Exclusion criteria:

* The score of contralateral knee pain (if present) >3.0 NRS at screening visit.
* Ipsilateral hip OA.
* Participant with systemic corticosteroids within 12 weeks prior to screening visit.
* Participant with injection of IA corticosteroids in the target knee joint within 26 weeks prior to screening visit.
* Concurrent chronic pain conditions with pain score >3.0 NRS at screening, or peripheral or central neuropathy that may affect sensation of the target knee area, including but not limited to back pain, hip pain, disc herniation, sciatica, diabetic neuropathy, post-stroke pain or fibromyalgia.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (21):
- China (21):
  - Investigational Site Number 1560001, Beijing
  - Investigational Site Number 1560005, Beijing
  - Investigational Site Number 1560020, Beijing
  - Investigational Site Number 1560009, Beijing
  - Investigational Site Number 1560012, Changchun
  - Investigational Site Number 1560013, Changsha
  - Investigational Site Number 1560023, Chengdu
  - Investigational Site Number 1560016, Guangzhou
  - Investigational Site Number 1560011, Hohhot
  - Investigational Site Number 1560017, Kunming
  - Investigational Site Number 1560019, Nanjing
  - Investigational Site Number 1560021, Nanjing
  - Investigational Site Number 1560007, Qingdao
  - Investigational Site Number 1560002, Shanghai
  - Investigational Site Number 1560003, Shanghai
  - Investigational Site Number 1560022, Shanghai
  - Investigational Site Number 1560018, Taiyuan
  - Investigational Site Number 1560010, Tianjin
  - Investigational Site Number 1560015, Tianjin
  - Investigational Site Number 1560006, Wuhan
  - Investigational Site Number 1560008, Wuxi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Ke Y, Jiang W, Xu Y, Chen Y, Zhang Q, Xue Q, Lin J, Ngai W, Nian G, Fazeli MS, Xie Y, Zhu Z. Efficacy and safety of a single intra-articular injection of 6 ml Hylan G-F 20 compared to placebo in Chinese patients with symptomatic knee osteoarthritis : C-SOUND study, a 26-week multicenter double-blind randomized placebo-controlled trial in China. BMC Musculoskelet Disord. 2021 May 8;22(1):428. doi: 10.1186/s12891-021-04252-2. PMID 33964907

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 21 sites in China from 21 August 2017 to 28 January 2019. A total of 524 participants were screened, of which, 84 participants were screen failures. Screen failures were mainly due to inclusion criteria not met.
Pre-assignment Details: A total of 440 participants were enrolled and randomized in the study. Assignment to arms was done centrally using an interactive voice response system/interactive web response system (IVRS/IWRS) in 1:1 ratio (Placebo: Hylan G-F 20).
Groups:
- Placebo: Participants received a single intra-articular (IA) injection of phosphate buffered saline on Day 1 and were observed for 26 weeks.
Period: Overall Study
Arm/Group | Placebo | Hylan G-F 20
Started | 220 | 220
Treated | 220 | 218
Completed | 219 | 212
Not Completed | 1 | 8
Not completed — Poor compliance to protocol | 0 | 1
Not completed — Withdraw before treatment | 1 | 5
Not completed — Randomized but not treated | 0 | 2

BASELINE CHARACTERISTICS:
Population: Analysis was performed on randomized population which consisted of all participants with a treatment kit number allocated and recorded in IVRS/IWRS database, and regardless of whether the treatment kit was used or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Hylan G-F 20 | Total
Number analyzed (Participants) | 220 | 220 | 440
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (7.8) | 61.5 (7.9) | 61.5 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172 | 170 | 342
  Male | 48 | 50 | 98
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 220 | 220 | 440
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) A1 Pain (Walking Pain) Subscale Score Over 26 Weeks
Description: The WOMAC Numerical Rating Scale (NRS) version 3.1 questionnaire was a self-administered, health status measure questionnaire of 24 questions comprising 3 subscales (joint pain, stiffness and physical function) for participants with Osteoarthritis (OA) of the knee. WOMAC A1 pain subscale (measure of pain during walking on a flat surface) was measured on 11-point (NRS) ranging from 0 (none) to 10 (extreme), where lower score represented no pain and higher score represented extreme pain.
Time Frame: From Baseline up to Week 26
Population: Analysis was performed on modified Intent-To-Treat (mITT) population which included all randomized and treated participants. Participants were analyzed in the treatment group to which they were randomized.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Hylan G-F 20
Number analyzed (Participants) | 220 | 218
score on a scale | -2.271 (0.110) | -2.146 (0.108)
Statistical Analysis 1: Comparison: Placebo vs Hylan G-F 20; Least-square (LS) means, standard errors (SE) were analyzed from repeated measures analysis of covariance (ANCOVA). The model included treatment groups (Hylan G-F 20 and placebo), site, visit and visit by treatment interaction, as well as the baseline WOMAC A1 score as a covariate); Test type: Superiority; p = 0.3610, ANCOVA — Threshold for significance at 0.05 level; Least-square (LS) means, standard errors (SE) were analyzed from repeated measures ANCOVA; LS Mean difference = 0.125, 95% CI 2-sided [-0.144 to 0.395], Standard Error of Mean 0.137

2. Secondary Outcome: Change From Baseline in 7-day Average WOMAC A1 Pain (Walking Pain) Subscale Score Over 26 Weeks
Description: The WOMAC NRS version 3.1 questionnaire was a self-administered, health status measure questionnaire of 24 questions comprising 3 subscales (joint pain, stiffness and physical function) for participants with OA of the knee. WOMAC A1 pain subscale (measure of pain during walking on a flat surface) was measured on 11-point (NRS) ranging from 0 (none) to 10 (extreme), where lower score represented no pain and higher score represented extreme pain. For 7-day average WOMAC A1, the baseline value was defined as the average of the WOMAC A1 scores recorded 7 days prior to the first investigational medicinal product (IMP) administration (WOMAC A1 score recorded on Day 1 included). The 7-day average WOMAC A1 was set as missing if 3 or more of the 7 WOMAC A1 scores were missing.
Time Frame: From Baseline up to Week 26
Population: Analysis was performed on mITT population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Hylan G-F 20
Number analyzed (Participants) | 220 | 218
score on a scale | -2.275 (0.108) | -2.176 (0.106)

3. Secondary Outcome: Change From Baseline in WOMAC A Score Over 26 Weeks
Description: The WOMAC NRS version 3.1 questionnaire was a self-administered, health status measure questionnaire of 24 questions comprising 3 subscales (joint pain, stiffness and physical function) for participants with OA of the knee. WOMAC A (5 items: measure of pain while walking, using stairs, at night while in bed, sitting or lying, and standing); each item was measured on 11-point (NRS) ranging from 0 (none) to 10 (extreme), where lower score represented no pain and higher score represented extreme pain. Total WOMAC A score was the sum of 5 item scores and ranges from 0 (none) to 50 (extreme); where lower score represented no pain and higher score represented extreme pain.
Time Frame: From Baseline up to Week 26
Population: Analysis was performed on mITT population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Hylan G-F 20
Number analyzed (Participants) | 220 | 218
score on a scale | -8.747 (0.491) | -8.621 (0.486)

4. Secondary Outcome: Change From Baseline in Patient Global Self-Assessment (PTGA) Score of Osteoarthritis Over 26 Weeks
Description: PTGA (self-assessment of target knee OA condition) was measured using an 11-point NRS ranging from 0 (best possible) to 10 (worst possible), where lower score represented best possible condition and higher score represented worst possible condition.
Time Frame: From Baseline up to Week 26
Population: Analysis was performed on mITT population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Hylan G-F 20
Number analyzed (Participants) | 220 | 218
score on a scale | -2.138 (0.104) | -2.144 (0.102)

5. Secondary Outcome: Change From Baseline in Clinical Observer Global Assessment (COGA) Score of Osteoarthritis Over 26 Weeks
Description: COGA was used by the physicians to perform a global assessment of the participant's target knee OA condition. The response was captured using the 11-point NRS pain intensity rating scale ranging from 0 (best possible) to 10 (worst possible) at the specified time points, where lower score represented best possible condition and higher score represented worst possible condition.
Time Frame: From Baseline up to Week 26
Population: Analysis was performed on mITT population.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Hylan G-F 20
Number analyzed (Participants) | 220 | 218
score on a scale | -2.145 (0.095) | -2.225 (0.094)

6. Secondary Outcome: Percentage of Positive WOMAC A1 Responder Over 26 Weeks
Description: WOMAC A1 responder were defined as >=2-point improvement from baseline in the WOMAC A1 NRS. The WOMAC NRS version 3.1 questionnaire was a self-administered, health status measure questionnaire of 24 questions comprising 3 subscales (joint pain, stiffness and physical function) for participants with OA of the knee. WOMAC A1 pain subscale (measure of pain during walking on a flat surface) was measured on 11-point (NRS) ranging from 0 (none) to 10 (extreme), where lower score represented no pain and higher score represented extreme pain.
Time Frame: Week 4, Week 8, Week 12, Week 16, Week 20 and Week 26
Population: Analysis was performed on mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Hylan G-F 20
Number analyzed (Participants) | 220 | 218
percentage of participants
  Week 4 | 58.6 | 53.2
  Week 8 | 65.0 | 62.4
  Week 12 | 66.4 | 62.8
  Week 16 | 69.1 | 63.3
  Week 20 | 65.0 | 66.5
  Week 26 | 68.2 | 67.0

7. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Adverse Event (AE) was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily had a causal relationship with the treatment. TEAEs were defined as AEs that developed, worsened (according to the Investigator opinion), or became serious during the on-treatment period (time from the injection of IMP up to Week 26 follow-up visit).
Time Frame: From Baseline up to Week 26
Population: Analysis was performed on safety population which included randomized participants who received at least 1 injection or part of an injection of Hylan G-F 20 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Hylan G-F 20
Number analyzed (Participants) | 220 | 218
Participants | 142 | 134

ADVERSE EVENTS:
Time Frame: AE data was collected from the time of the injection of IMP up to Week 26 follow-up visit.
Description: Reported AEs are TEAEs that developed, worsened, or became serious during the treatment period (time from the injection of IMP up to Week 26 follow-up visit). Analysis was performed on safety population.
Arm/Group | Placebo | Hylan G-F 20
All-Cause Mortality (participants affected / at risk) | 0/220 | 0/218
Serious Adverse Events (participants affected / at risk) | 10/220 | 14/218
Other Adverse Events (participants affected / at risk) | 66/220 | 75/218
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=220) | Hylan G-F 20 (N=218)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis B (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cerebral Infarction (Nervous system disorders) | 1 (1) | 1 (1)
Lacunar Infarction (Nervous system disorders) | 0 (0) | 1 (1)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 2 (2)
Abdominal Adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Uterine Polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Joint Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament Sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=220) | Hylan G-F 20 (N=218)
Nasopharyngitis (Infections and infestations) | 12 (18) | 13 (14)
Upper Respiratory Tract Infection (Infections and infestations) | 30 (40) | 28 (31)
Toothache (Gastrointestinal disorders) | 8 (9) | 11 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 (29) | 26 (35)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 4 (5) | 16 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2017-02-17): https://cdn.clinicaltrials.gov/large-docs/69/NCT03190369/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/69/NCT03190369/SAP_001.pdf